CLINICAL TRIAL: NCT06111820
Title: Evaluation of Training Curriculum and Service of Improving Access to Community Therapies
Acronym: iACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mind Mental Health Hong Kong Limited (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHK/2023/R01-PWP
Record Dates: First submitted 2023-10-10; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Depression; Anxiety; Mental Health Issue; Stress; Distress, Emotional
Keywords: Psychotherapies; Psychological therapies; Evaluation; Improving access; Community therapy; Community therapies; Low-intensity; Acceptance and Commitment Therapy; ACT
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iACT service users (Experimental): All participants enrolled in the programme will participate in the iACT service referring to the aforementioned details.
  Interventions: Behavioral: Improving Access to Community Therapies (iACT)

INTERVENTIONS:
Behavioral: Improving Access to Community Therapies (iACT) — The Low-intensity Acceptance and Commitment Therapy (LIACT) protocol is based on the empirically supported Acceptance and Commitment Therapy (ACT), and is designed by registered clinical psychologists with consultation from local ACT experts from the Association of Contextual and Behavioural Science (Hong Kong Chapter). The LIACT protocol is also piloted and revised by clinical psychologists to ensure its adaptability to local situations. For individual guided self-help LIACT service, an intake assessment will be conducted to assess the presenting problem of the participants at pre-treatment to ensure the suitability to receive LIACT service. Participants will be given the LIACT self-help workbook collaboratively with a Psychological Wellbeing Practitioner (PWP). Between each session, clients will read through the workbook and complete the exercises suggested in the workbook. In subsequent sessions, PWP will guide clients to overcome the difficulties in performing the LIACT exercises.
  Other Names: Manualised Acceptance and Commitment Therapy (ACT); Low-intensity Acceptance and Commitment Therapy (LIACT)

SUMMARY:
The current study aims to conduct a comprehensive evaluation of a training curriculum designed for teaching low-intensity psychological interventions to bachelor's degree holders, specifically focusing on principles of Acceptance and Commitment Therapy (ACT) and its intervention effectiveness. This evaluation is divided into two integral parts.

In the first part, the curriculum, which encompasses a 120-hour intensive teaching block followed by a nine-month placement, will be evaluated. To assess the trainees' competencies in applying the principles of ACT, a series of role-play examinations will be administered at various time points, including pre-training, pre-placement, mid-placement, and end-of-placement. Focus groups will be conducted.

The second part of the evaluation is to examine the outcomes of low-intensity psychological interventions, delivered by the trainees, targeting adult individuals screened with mild to severe symptoms of depression and anxiety. To achieve this, a series of questionnaires will be administered at several stages: pre-intervention, during each session, and at a three-month follow-up. Outcome measures will include the assessment of depressive and anxiety symptom severity, quality of life, functional impairment, therapeutic alliance, and the level of experiential avoidance. Individual exit interviews and focus groups will be conducted.

The aim of the study:

1. To evaluate the effectiveness of the training program
2. To evaluate the effectiveness of the low-intensity psychological intervention based on the Acceptance and Commitment Therapy (ACT) principle

Hypotheses:

It is hypothesised that the competency level of the training participants will increase after the intensive training block and the placement. It is also hypothesised that after receiving the low-intensity psychological intervention based on the ACT principle, the depression and anxiety scores, functioning impairment, and experiential avoidance level will reduce, and quality of life and therapeutic relationship will improve.

DETAILED DESCRIPTION:
'Training Participants': Participants from the Psychological Wellbeing Practitioners (PWPs) Programme will be invited to participate in the research. The PWPs are bachelors. Degree holders will undergo 120 hours of intensive training block, followed by a 9-month placement to practise the learnt skills. Given therapist competency will be part of the program, this research will request the participants to consent to the use of the data collected in the program.

'Service Participants': Individuals with depression or anxiety symptoms will be sampled in this study. Participants will be recruited from the placement organisations and promotions on social media, web pages, and at mental health centres. The sample size is estimated to be 300 individuals for initial screening for LIACT-guided self-help services.

Research design:

For training evaluation, given the current training programme already consists of a therapist competency assessment to ensure the quality of the training participants. Recorded role-play videos will be rated the ACT therapist competency by trained psychologists at pre-training, post-training block, mid-placement and post-placement. A consent form will be sent to the training participant to authorise the use of data for analysis.

Repeated measures design will be adopted for this study. Individual guided self-help LIACT service, eligible participants will receive 6-8 sessions of guided self-help LIACT over three to four months. Clinical outcomes (depression and anxiety levels) will be measured at every session, it will take around 5 minutes to complete these two routine outcome measures. Other primary and secondary outcome measures, including functioning impairment, quality of life, psychological flexibility, experiential avoidance, absenteeism, and therapeutic alliance will be at 3 time points, namely pre-treatment, post-treatment (at the end of the last session) and 3-month follow-up. Participants will take around 30 minutes to complete the full package of assessments. These outcome variables will be additionally measured after each session to avoid missing data if participants drop out. The recovery rate and reliable improvement rate will also be used as indicators to evaluate the efficacy of LIACT. Focus groups will be conducted on participants who drop out and complete the programme to understand their experience and journey.

Curriculum The LIACT training curriculum is designed by registered clinical psychologists with consultation from local ACT experts from the Association of Contextual and Behavioural Science (Hong Kong Chapter). There are 5 modules in the intensive training block including introduction, professional and ethics issues, application of ACT low-intensity intervention, troubleshooting and preparation for clinical placement. The LIACT protocol is also piloted and revised by clinical psychologists to ensure its adaptability to local situations. After 120- hour intensive training, the training participants will attend a role play exam to ensure their competency to proceed with the 9-month placement. During the 9-month placement, each PWP is expected to see at least 15 direct service beneficiaries to provide LIACT. During this supervision will be provided regularly to ensure the quality of service delivery and risk management. There will be a mid-placement review and final placement review, and the training participants will submit audio recordings for supervisors to rate for their competence.

A focus group will be conducted for the training participants to understand their learning experience.

Treatment Guided self-help LIACT will be provided to eligible participants. For individual guided self-help LIACT service, an intake assessment will be conducted to assess the presenting problem of the participants at pre-treatment to ensure the suitability to receive LIACT service. Participants will be given the LIACT self-help workbook collaboratively with a PWP. Between each session, clients will read through the workbook and complete the exercises suggested in the workbook. In subsequent sessions, PWP will guide clients to overcome the difficulties in performing the LIACT exercises.

Therapists PWPs will be responsible for providing LIACT to the participants. PWPs have completed a 120-hour intensive training and pass the role play examination prior to placement provision. The training was provided by experienced clinical psychologists and counsellors. Moreover, PWPs are under regular supervision by clinical psychologists, experienced counsellors, or social workers with extensive ACT training.

ELIGIBILITY:
Inclusion Criteria:

18-65 years old adults with any of the following problem(s):

* Anxiety problem (including social, generalised, health anxiety, work anxiety)
* Mild to moderate depression
* Other emotional challenges including (but not limited to) low self esteem, perfectionism, mild anger issues, interpersonal or relational challenges, low motivation, lack of purpose, numbness.

Exclusion Criteria:

Adults with the following features/ presentations are not eligible for the PWP programme and should automatically lead to an onward referral:

* High severity on the depressive score (PHQ9 >= 20)
* High or imminent risk (according to scores on PHQ9 question no. 9 and information emerging at triage assessment, including indication of plan and action or the lack of protective factor)

Individuals with any of the following diagnoses or situations are also excluded:

* Obsessive-compulsive disorder
* Post-traumatic stress disorder
* Bipolar disorder
* Schizophrenia and other psychotic disorders
* Dissociative disorders
* Personality disorders
* Eating disorders
* Gender dysphoria
* Paraphilic disorders
* Anger issues as primary presenting concern (without anxiety or depression)
* Sleep issues as primary presenting concern (without anxiety or depression)
* Substance-related disorders
* History of trauma or abuse that is considered highly relevant to the current presenting problem they are seeking support for
* Planned changes to psychotropic medication during the period of PWP intervention
* Currently receiving regular psychological counselling or support from another practitioner.
* Diagnosis of a learning disability, cognitive impairment or neurodevelopmental condition that would impair their ability to engage with a structured, manualised intervention (e.g. untreated ADHD or moderate-severe brain injury)
* Clients with unstable or unsafe home environments (e.g. domestic abuse)
* Clear safeguarding concerns requiring multi-agency support (e.g. concerns about child abuse or neglect)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2022-05-22 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
ACT Fidelity Measure (ACT-FM) | Pre-training, post-training (2nd month), during mid-placement review (6th month), and during end-of-placement (11th month)
  This measure is intended to be used by clinicians who are experienced in ACT to rate the competencies of their therapists. It can be used to measure fidelity to ACT in a variety of contexts (e.g. as a tool to evaluate your own or another clinician's practice, or as a research tool). The items capture four key areas within ACT: Therapist Stance, Open Response Style, Aware Response Style and Engaged Response Style. Scoring is broken down into two subgroups - ACT Consistency Score and ACT Inconsistency Score.
Enhancing Assessment of Common Therapeutic Factors (ENACT) scale | Pre-training, post-training (2nd month), during mid-placement review (6th month), and during end-of-placement (11th month)
  The ENACT scale is a measurement tool used in clinical psychology and psychotherapy research to assess common therapeutic factors in therapeutic interventions. It measures elements such as the therapeutic alliance, empathy, collaboration, goal consensus, and client involvement. The scale consists of self-report items rated on a Likert scale, providing a quantitative assessment of these factors. It helps therapists and researchers understand the therapeutic process, identify areas for improvement, and explore the relationship between common therapeutic factors and treatment outcomes. Score: 18-54, the higher the more competent in general counselling.
Patient Health Questionnaire-9 (PHQ-9) | 1) During clients' enrolment 2) before intake interview (week 0) 3) weekly from session 1 to session 6, and 4) before follow-up (week 12).
  The PHQ-9 questions are based on diagnostic criteria of depression from DSM-IV and ask about the patient's experience in the last 2 weeks. Questions are about the level of interest in doing things, feeling down or depressed, difficulty with sleeping, energy levels, eating habits, self-perception, ability to concentrate, speed of functioning and thoughts of suicide. Score: 0-27, the higher the more depressed.
Generalised Anxiety Disorder Assessment (GAD-7) | During clients' enrolment 2) before intake interview (week 0), weekly from session 1 to session 6, and before follow-up (week 12).
  The Generalised Anxiety Disorder 7 (GAD-7) is a self-reported questionnaire for screening and severity measuring of generalised anxiety disorder (GAD). Score: 0-21, the higher the more anxious.
The Work and Social Adjustment Scale (WSAS) | Before intake interview (week 0), after session 6 (week 6), and before follow-up (week 12).
  WSAS is a 5-item, self-report measure of impairment in functioning. It assesses the impact of a person's mental health difficulties on their ability to function in terms of work, home management, social leisure, private leisure and personal or family relationships. Score: 0-40, the higher the more severe the impairment.
The World Health Organisation - Five Well-Being Index (WHO-5) | Before intake interview (week 0), after session 6 (week 6), and before follow-up (week 12).
  The WHO-5 is a questionnaire that measures current mental well-being (time frame the previous two weeks)." Originally developed to assess both positive and negative well-being, this five question version use only positively phrased questions to avoid symptom-related language. Score: 0-25, the higher the better well-being.

SECONDARY OUTCOMES:
Work Productivity and Activity Impairment Questionnaire: General Health V2.0 (WPAI:GH) | Before intake interview (week 0), after session 6 (week 6), and before follow-up (week 12).
  WPAI is a 6-item self-report questionnaire used to assess the impact of health conditions on work productivity and daily activities. It consists of a series of questions that inquire about different aspects of work productivity and activity impairment. It assesses absenteeism (time missed from work due to health issues), presenteeism (reduced productivity while at work due to health issues), overall work productivity impairment, and activity impairment in non-work-related activities. Score: 0-20, the higher the more severe. And the higher the number of hours reported, the more occupationally impaired.
Brief Revised Working Alliance Inventory (BR-WAI) | Before session 1 (week 1), session 4 (week 4) and session 6 (week 6).
  BR-WAI is a 12-item self-report measure of the therapeutic alliance that assesses three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond. Score: 12-60. The higher the stronger the therapeutic alliance.
Brief Experiential Avoidance Questionnaire (BEAQ) | Before intake interview (week 0), after session 6 (week 6), and before follow-up (week 12).
  The 15-item self-report measure assesses experiential avoidance or the avoidance of uncomfortable or distressing thoughts and emotions. Score: 6-90. The higher the more avoidance.
Acceptance and Action Questionnaire II (AAQ-II) | Before intake interview (week 0), after session 6 (week 6), and before follow-up (week 12).
  This 7-item scale is the most widely used measure of psychological flexibility. Score: 7-49, the higher the less psychologically flexible.

CONTACTS AND LOCATIONS:
Overall Officials: Candice LYM Powell, Principal Investigator — Mind Mental Health Hong Kong Limited; Patrick WL Leung, Principal Investigator — Chinese University of Hong Kong
Locations (21):
- China (21):
  - Aberdeen Kai-fong Welfare Association Services Centre, Hong Kong
  - Baptist Oi Kwan Social Service, Hong Kong
  - Cedar Communications Ltd, Hong Kong
  - Central Health, Hong Kong
  - Central Minds, Hong Kong
  - Fu Hong Society, Hong Kong
  - HKU Lap-Chee College, Hong Kong
  - HKUSPACE PLK Stanley Ho Community College, Hong Kong
  - Hong Kong Physically Handicapped and Able-Bodied (PHAB) Association, Hong Kong
  - KUNST EXA Academy, Hong Kong
  - LU Institute of Further Education, Hong Kong
  - Mind Mental Health Hong Kong Limited, Hong Kong
  - MINDSET, Hong Kong
  - PathFinders Hong Kong, Hong Kong
  - Run HK, Hong Kong
  - Society for Community Organisation (SoCO), Hong Kong
  - St. John's Cathedral Counselling Service, Hong Kong
  - The Hong Kong Federation of Youth Groups, Hong Kong
  - The Mental Health Association of Hong Kong, Hong Kong
  - WYNG Foundation, Hong Kong
  - Yuen Long Town Hall, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alonso J, Angermeyer MC, Bernert S, Bruffaerts R, Brugha TS, Bryson H, de Girolamo G, Graaf R, Demyttenaere K, Gasquet I, Haro JM, Katz SJ, Kessler RC, Kovess V, Lepine JP, Ormel J, Polidori G, Russo LJ, Vilagut G, Almansa J, Arbabzadeh-Bouchez S, Autonell J, Bernal M, Buist-Bouwman MA, Codony M, Domingo-Salvany A, Ferrer M, Joo SS, Martinez-Alonso M, Matschinger H, Mazzi F, Morgan Z, Morosini P, Palacin C, Romera B, Taub N, Vollebergh WA; ESEMeD/MHEDEA 2000 Investigators, European Study of the Epidemiology of Mental Disorders (ESEMeD) Project. Disability and quality of life impact of mental disorders in Europe: results from the European Study of the Epidemiology of Mental Disorders (ESEMeD) project. Acta Psychiatr Scand Suppl. 2004;(420):38-46. doi: 10.1111/j.1600-0047.2004.00329.x. PMID 15128386
- [Background] Antony, M. M., Bieling, P. J., Cox, B. J., Enns, M. W., & Swinson, R. P. (1998). Psychometric Properties of the 42-Item and 21-Item Versions of the Depression Anxiety Stress Scales in Clinical Groups and a Community Sample. Psychological assessment, 10(2), 176-181.
- [Background] Bai Z, Luo S, Zhang L, Wu S, Chi I. Acceptance and Commitment Therapy (ACT) to reduce depression: A systematic review and meta-analysis. J Affect Disord. 2020 Jan 1;260:728-737. doi: 10.1016/j.jad.2019.09.040. Epub 2019 Sep 10. PMID 31563072
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Belanger L, Savard J, Morin CM. Clinical management of insomnia using cognitive therapy. Behav Sleep Med. 2006;4(3):179-198. doi: 10.1207/s15402010bsm0403_4. PMID 16879081
- [Background] Chung KF, Ho FY, Yeung WF. Psychometric Comparison of the Full and Abbreviated Versions of the Dysfunctional Beliefs and Attitudes about Sleep Scale. J Clin Sleep Med. 2016 Jun 15;12(6):821-8. doi: 10.5664/jcsm.5878. PMID 26857054
- [Background] Clark DM. Implementing NICE guidelines for the psychological treatment of depression and anxiety disorders: the IAPT experience. Int Rev Psychiatry. 2011 Aug;23(4):318-27. doi: 10.3109/09540261.2011.606803. PMID 22026487
- [Background] Clark DM, Layard R, Smithies R, Richards DA, Suckling R, Wright B. Improving access to psychological therapy: Initial evaluation of two UK demonstration sites. Behav Res Ther. 2009 Nov;47(11):910-20. doi: 10.1016/j.brat.2009.07.010. Epub 2009 Jul 14. PMID 19647230
- [Background] Cuijpers P, Donker T, van Straten A, Li J, Andersson G. Is guided self-help as effective as face-to-face psychotherapy for depression and anxiety disorders? A systematic review and meta-analysis of comparative outcome studies. Psychol Med. 2010 Dec;40(12):1943-57. doi: 10.1017/S0033291710000772. Epub 2010 Apr 21. PMID 20406528
- [Background] Espie CA, Inglis SJ, Harvey L, Tessier S. Insomniacs' attributions. psychometric properties of the Dysfunctional Beliefs and Attitudes about Sleep Scale and the Sleep Disturbance Questionnaire. J Psychosom Res. 2000 Feb;48(2):141-8. doi: 10.1016/s0022-3999(99)00090-2. PMID 10719130
- [Background] Gyani A, Shafran R, Layard R, Clark DM. Enhancing recovery rates: lessons from year one of IAPT. Behav Res Ther. 2013 Sep;51(9):597-606. doi: 10.1016/j.brat.2013.06.004. Epub 2013 Jul 4. PMID 23872702
- [Background] Haller H, Breilmann P, Schroter M, Dobos G, Cramer H. A systematic review and meta-analysis of acceptance- and mindfulness-based interventions for DSM-5 anxiety disorders. Sci Rep. 2021 Oct 14;11(1):20385. doi: 10.1038/s41598-021-99882-w. PMID 34650179
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Janssen MF, Pickard AS, Golicki D, Gudex C, Niewada M, Scalone L, Swinburn P, Busschbach J. Measurement properties of the EQ-5D-5L compared to the EQ-5D-3L across eight patient groups: a multi-country study. Qual Life Res. 2013 Sep;22(7):1717-27. doi: 10.1007/s11136-012-0322-4. Epub 2012 Nov 25. PMID 23184421
- [Background] Jacobson NS, Truax P. Clinical significance: a statistical approach to defining meaningful change in psychotherapy research. J Consult Clin Psychol. 1991 Feb;59(1):12-9. doi: 10.1037//0022-006x.59.1.12. PMID 2002127
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837
- [Background] Kyllönen, H. M., Muotka, J., Puolakanaho, A., Astikainen, P., Keinonen, K., & Lappalainen, R. (2018). A brief acceptance and commitment therapy intervention for depression: A randomized controlled trial with 3-year follow-up for the intervention group. Journal of contextual behavioral science, 10, 55-63.
- [Background] Kroenke, K., & Spitzer, R. L. (2002). The PHQ-9: A New Depression Diagnostic and Severity Measure. Psychiatric annals, 32(9), 509-515. doi:10.3928/0048-5713-20020901-06
- [Background] Lam LC, Wong CS, Wang MJ, Chan WC, Chen EY, Ng RM, Hung SF, Cheung EF, Sham PC, Chiu HF, Lam M, Chang WC, Lee EH, Chiang TP, Lau JT, van Os J, Lewis G, Bebbington P. Prevalence, psychosocial correlates and service utilization of depressive and anxiety disorders in Hong Kong: the Hong Kong Mental Morbidity Survey (HKMMS). Soc Psychiatry Psychiatr Epidemiol. 2015 Sep;50(9):1379-88. doi: 10.1007/s00127-015-1014-5. Epub 2015 Feb 8. PMID 25660760
- [Background] Lim D, Sanderson K, Andrews G. Lost productivity among full-time workers with mental disorders. J Ment Health Policy Econ. 2000 Sep 1;3(3):139-146. doi: 10.1002/mhp.93. PMID 11967449
- [Background] Lovibond PF, Rapee RM. The representation of feared outcomes. Behav Res Ther. 1993 Jul;31(6):595-608. doi: 10.1016/0005-7967(93)90111-7. PMID 8347118
- [Background] Meyer TJ, Miller ML, Metzger RL, Borkovec TD. Development and validation of the Penn State Worry Questionnaire. Behav Res Ther. 1990;28(6):487-95. doi: 10.1016/0005-7967(90)90135-6. PMID 2076086
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Background] School of Health and Related Research (ScHARR), University of Sheffield. Clinical Guidelines for the Management of Anxiety: Management of Anxiety (Panic Disorder, with or without Agoraphobia, and Generalised Anxiety Disorder) in Adults in Primary, Secondary and Community Care [Internet]. London: National Collaborating Centre for Primary Care (UK); 2004 Dec. Available from http://www.ncbi.nlm.nih.gov/books/NBK45834/ PMID 20945576
- [Background] National Institute for Health and Clinical Excellence [NICE]. (2009). Depression: treatment and management of depression in adults, including adults with a chronic physical health problem: NICE.
- [Background] National Institute for Health and Care Excellence [NICE]. (2011, 05 25). Retrieved 06 15, 2022, from Common mental health problems: identification and pathways to care: https://www.nice.org.uk/guidance/cg123/chapter/Recommendations
- [Background] Ng SS, Lo AW, Leung TK, Chan FS, Wong AT, Lam RW, Tsang DK. Translation and validation of the Chinese version of the short Warwick-Edinburgh Mental Well-being Scale for patients with mental illness in Hong Kong. East Asian Arch Psychiatry. 2014 Mar;24(1):3-9. PMID 24676481
- [Background] Richards DA, Suckling R. Improving access to psychological therapies: phase IV prospective cohort study. Br J Clin Psychol. 2009 Nov;48(Pt 4):377-96. doi: 10.1348/014466509X405178. Epub 2009 Feb 9. PMID 19208291
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Stewart-Brown S, Tennant A, Tennant R, Platt S, Parkinson J, Weich S. Internal construct validity of the Warwick-Edinburgh Mental Well-being Scale (WEMWBS): a Rasch analysis using data from the Scottish Health Education Population Survey. Health Qual Life Outcomes. 2009 Feb 19;7:15. doi: 10.1186/1477-7525-7-15. PMID 19228398
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] Wang K, Shi HS, Geng FL, Zou LQ, Tan SP, Wang Y, Neumann DL, Shum DH, Chan RC. Cross-cultural validation of the Depression Anxiety Stress Scale-21 in China. Psychol Assess. 2016 May;28(5):e88-e100. doi: 10.1037/pas0000207. Epub 2015 Nov 30. PMID 26619091
- [Background] Wang W, Bian Q, Zhao Y, Li X, Wang W, Du J, Zhang G, Zhou Q, Zhao M. Reliability and validity of the Chinese version of the Patient Health Questionnaire (PHQ-9) in the general population. Gen Hosp Psychiatry. 2014 Sep-Oct;36(5):539-44. doi: 10.1016/j.genhosppsych.2014.05.021. Epub 2014 Jun 6. PMID 25023953
- [Background] White, J. (2000). Treating anxiety and stress : a group psycho-educational approach using brief CBT. Chichester ; New York: Wiley.
- [Background] Whiteford HA, Degenhardt L, Rehm J, Baxter AJ, Ferrari AJ, Erskine HE, Charlson FJ, Norman RE, Flaxman AD, Johns N, Burstein R, Murray CJ, Vos T. Global burden of disease attributable to mental and substance use disorders: findings from the Global Burden of Disease Study 2010. Lancet. 2013 Nov 9;382(9904):1575-86. doi: 10.1016/S0140-6736(13)61611-6. Epub 2013 Aug 29. PMID 23993280
- [Background] Williams M, Honan C, Skromanis S, Sanderson B, Matthews AJ. Psychological Outcomes and Mechanisms of Mindfulness-Based Training for Generalised Anxiety Disorder: A Systematic Review and Meta-Analysis. Curr Psychol. 2023 May 11:1-23. doi: 10.1007/s12144-023-04695-x. Online ahead of print. PMID 37359641
- [Background] World Health Organization. (2017). Depression and other common mental disorders: global health estimates. World Health Organization.
- [Background] Yu DS. Insomnia Severity Index: psychometric properties with Chinese community-dwelling older people. J Adv Nurs. 2010 Oct;66(10):2350-9. doi: 10.1111/j.1365-2648.2010.05394.x. Epub 2010 Aug 16. PMID 20722803
- [Background] Zhong J, Wang C, Li J, Liu J. Penn State Worry Questionnaire: structure and psychometric properties of the Chinese version. J Zhejiang Univ Sci B. 2009 Mar;10(3):211-8. doi: 10.1631/jzus.B0820189. PMID 19283876
- See also: Enrolment website of the iACT intervention services. — https://www.iact.hk/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/20/NCT06111820/Prot_SAP_000.pdf